CLINICAL TRIAL: NCT03783780
Title: Desaturation Validation of INVSENSOR00031
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-19564
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Results first posted 2019-07-02 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- INVSENSOR00031 (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00031 sensor during motion and non-motion.
  Interventions: Device: INVSENSOR00031

INTERVENTIONS:
Device: INVSENSOR00031 — Noninvasive pulse oximeter sensor

SUMMARY:
This study is designed to compare the accuracy of a noninvasive measurement of oxygen saturation compared to reference values obtained by a laboratory blood gas analyzer. Arterial blood samples will be collected from healthy adult subjects while undergoing a desaturation procedure wherein the concentration of oxygen inhaled is slowly reduced until the subject's arterial oxygen concentration is approximately 70%. During the desaturation, the subject's hand and arm without the arterial line will be subjected to motion at various times during the study. The subject will then be returned to breathing room air.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-50 years of age.
* Subject weighs a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
* Hemoglobin value is greater than or equal to 11 g/dL.
* Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
* Carbon monoxide (CO) value ≤ 2.0% fractional carboxyhemoglobin (FCOHb)
* Subject has a physical status of ASA I or II (American Society of Anesthesiology Class I; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease) as it applies to the systemic disease portion of the classification.
* Systolic Blood Pressure ≤ 140 mmHg and Diastolic Blood Pressure ≤ 90 mmHg.
* Subject is able to read and communicate in English and understands the study and risks involved.

Exclusion Criteria:

* Subject is pregnant.
* Subject smokes (smoking includes e-cigarette use).
* Subject has a BMI > 35 and has been classified as morbidly obese or at an increased risk for participation by a medical professional.
* Subject has a history of fainting (vasovagal), blacking out or losing consciousness during or after blood draw, or has a fear of blood draws.
* Subject has open wounds, inflamed tattoos or piercings, or any visible healing wounds that a medical professional renders them at an increased risk for participation.*
* Subject experiences frequent or severe headaches and/or migraine headaches.
* Subject has known drug or alcohol abuse and/or use of recreational drugs.
* Subject has experienced a concussion or head injury with loss of consciousness within the last 12 months.
* Subject has any chronic bleeding disorders (i.e. hemophilia).
* Subject has any history of a stroke, myocardial infarction, seizures or heart attack.
* Subject has any cancer or history of cancer (not including skin cancer).*
* Subject has any cardiac dysrhythmia(s) (i.e. atrial fibrillation) and has not received clearance by their physician to participate.
* Subject has a known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder, Multiple Sclerosis, Huntington's Disease) that interferes with the subject's level of consciousness.
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
* Subject who has taken anticoagulant medication within the last 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDS)).
* Subject has taken opioid pain medication 24 hours before the study.
* Subject has any type of infectious disease (i.e. Hepatitis, HIV, Tuberculosis, Flu, Malaria, Measles, etc.)
* Subject is taking medications known to treat any type of infectious disease.
* Subject has either signs or history of peripheral ischemia.
* Subject has had invasive surgery within the past year- including but not limited to major dental surgery*, appendix*, plastic surgery*.
* Subject has had invasive surgery within the past year- including but not limited to gallbladder, heart, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, major ears, nose and throat (ENT) surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
* Subject has donated blood within the past 4 weeks.
* Subject has symptoms of congestion, head colds, flu or other illnesses.
* Subject experiences claustrophobia or has generalized anxiety disorder.
* Subject has been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the last 12 months.
* Subject has chronic unresolved asthma, lung disease or respiratory disease.
* Subject is allergic to lidocaine, latex, adhesives, or plastic.
* Subject has heart conditions, insulin-dependent Diabetes or uncontrolled hypertension.
* Subject has given vaginal delivery, had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the last 6 months.
* Subject intends to participate in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle) or exercise (working out, riding a bike, riding a skate board etc.), or any activity that will put additional stress on the wrist within 24 hours of the study.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00031
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawn prior to completion | 1

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00031
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants] — Population: One subject was withdrawn prior to completing study procedures.
  Participants
    number analyzed (Participants) | 20
    <=18 years | 0
    Between 18 and 65 years | 20
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject was withdrawn prior to completing study procedures.
  Participants
    number analyzed (Participants) | 20
    Female | 11
    Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One subject was withdrawn prior to completion of study procedures.
  Participants
    White: number analyzed (Participants) | 20
    White | 10
    Hispanic: number analyzed (Participants) | 20
    Hispanic | 5
    Asian or Pacific Islander: number analyzed (Participants) | 20
    Asian or Pacific Islander | 2
    African American: number analyzed (Participants) | 20
    African American | 3
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation (SpO2) Accuracy of Sensor by Arms Calculation During Non-motion
Description: Performance of the sensors will be determined by comparing the noninvasive oxygen saturation measurement (SpO2) of the pulse oximeter sensors to the arterial oxygen saturation (SaO2) value obtained from a reference blood sample and calculating the Arithmetic root mean square (ARMS) value during non-motion.
Time Frame: 1-5 hours
Population: Only ten subjects, out of the 20 who participated in the study, underwent testing for this non-motion outcome measure.
Measure: Number; unit: % of oxygen saturated hemoglobin
Groups:
- INVSENSOR00031: All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00031 sensor.
Arm/Group | INVSENSOR00031
Number analyzed (Participants) | 10
% of oxygen saturated hemoglobin | 1.33

2. Secondary Outcome: Oxygen Saturation (SpO2) Accuracy of Sensor by Arms Calculation During Motion
Description: Performance of the sensors will be determined by comparing the noninvasive oxygen saturation measurement (SpO2) of the pulse oximeter sensors to the arterial oxygen saturation (SaO2) value obtained from a reference blood sample and calculating the Arithmetic root mean square (ARMS) value during motion.
Time Frame: 1-5 hours
Population: Ten subjects were excluded from data analysis from this outcome measure due to insufficient training of the study staff on the motion testing procedure.
Measure: Number; unit: % of oxygen saturated hemoglobin
Arm/Group | INVSENSOR00031
Number analyzed (Participants) | 10
% of oxygen saturated hemoglobin | 2.16

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | INVSENSOR00031
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INVSENSOR00031 (N=21)
Scraped skin (Injury, poisoning and procedural complications) | 1 — Subjects skin was scraped with scissors, no visual abrasion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT03783780/Prot_SAP_000.pdf